CLINICAL TRIAL: NCT00942877
Title: Phase II Study of Cediranib (AZD2171) in Patients With Alveolar Soft Part Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 090192; 09-C-0192
Record Dates: First submitted 2009-07-18; First posted 2009-07-21 (Estimated); Results first posted 2021-04-27 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Sarcoma, Alveolar Soft Part
Keywords: VEGF; Antiangiogenesis; Tyrosine Kinase Inhibitor; Advanced Cancer; Alveolar Soft Part Sarcoma; Sarcoma
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Sarcoma | interventions — cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cediranib (AZD2171) Treatment (Experimental): Adult participants will be treated with 30 mg by mouth once a day for 28 days (28-day cycles).
  Pediatric participants (<16 years old) will be treated with 12 mg/m^2/day once a day for 28 days (28-day cycles).
  Interventions: Drug: AZD2171

INTERVENTIONS:
Drug: AZD2171 — Cediranib (AZD2171), a vascular endothelial growth factor (VEGF)/KIT tyrosine kinase inhibitor, has demonstrated antitumor activity in early phase clinical trials in adult and pediatric patients with Alveolar Soft Part Sarcoma (ASPS).
  Other Names: Cediranib

SUMMARY:
Background:

* Alveolar soft part sarcoma is a type of cancer that develops in tissues that connect, support, or surround other organs in the body. It relies heavily on new blood vessels to grow and spread through the body. There is no effective systemic treatment for patients with alveolar soft part sarcoma.
* The drug AZD2171 (cediranib) is an experimental drug, not yet approved by the Food and Drug Administration. The drug blocks the creation of new blood vessels. The drug has had initial clinical trials, and researchers are interested in determining whether cediranib is effective in inhibiting tumor growth in individuals who have alveolar soft part sarcoma.

Objectives:

- To find out whether AZD2171 works in patients who have alveolar soft part sarcoma.

Eligibility:

- Individuals 18 years of age and older who have been diagnosed with alveolar soft part sarcoma.

Design:

* After an initial screening visit, patients will take AZD2171 by mouth once a day, every day for the duration of the study. The treatment will be given in 28-day cycles.
* Patients will keep a study diary to record the doses taken, any missed doses, and any side effects.
* Patients will have the following tests and procedures during the treatment period: clinic visit with physical examination every 2 weeks during cycles 1 and 2, then at the start of each subsequent cycle, regular blood pressure monitoring, blood and urine tests, heart function tests, imagining scans to evaluate tumor size and response to the treatment, and possible tumor biopsy.

DETAILED DESCRIPTION:
Background:

Alveolar soft part sarcoma (ASPS) is a rare, highly vascular tumor accounting for less than 1% of soft tissue sarcomas. There is no effective systemic treatment for patients with metastatic ASPS. Little is known with regards to relevant molecular markers as potential therapeutic targets. Cediranib (AZD2171), a vascular endothelial growth factor (VEGF)/KIT tyrosine kinase inhibitor, has recently demonstrated antitumor activity in early phase clinical trials, which included 7 adult and 3 pediatric patients with ASPS.

Objectives:

Adult patients:

* To determine the response rate (Partial Response (PR) + Complete Response (CR)) of AZD2171 in adult patients with ASPS.
* To compare gene expression profiles between pre-treatment and post-treatment biopsy specimens.

Pediatric patients:

-To determine if pediatric patients with ASPS will experience at least a minimal response rate when treated with AZD2171

Eligibility:

Patients must have histologically or cytologically confirmed metastatic alveolar soft part sarcoma.

* Less than 16 years old. Body surface area (BSA) must be greater than or equal to 1.04 m^2 and subject must be able to swallow tablets.
* Adequate organ function.

Design:

Adult patients will be treated with AZD2171 at 30 mg by mouth once a day for 28 days (28-day cycles). Pediatric patients (< 16 years old) will be treated with 12 mg/m^2/day once a day for 28 day (28-day cycles).

Blood pressure will be monitored weekly for the first 2 cycles then every 2 weeks for the remainder of the study (unless patients have experienced elevated blood pressure requiring drug therapy).

Computed tomography (CT) scans will be performed at baseline and every 2 cycles for restaging during the first 18 months; after 18 and 36 months, restaging CT scans will be performed every 3 or 4 cycles, respectively.

The study will be conducted using an optimal two-stage design in both pediatric and adult patients. The portion in adults will rule out an unacceptably low 5% clinical response rate (PR+CR) in favor of a modestly high response rate of 25%. In pediatric patients, the study will rule out an unacceptably low 5% overall clinical response rate (CR + PR) in favor of a higher response rate of 35%.

Optional biopsies will be performed in adult patients only at baseline and after 3-5 days of treatment (Day 3 (D3)-Day 5 (D5)) to evaluate early drug effect. A third optional biopsy after completion of 4 weeks of therapy (between Cycle 1 Day 28 (C1D28) and Cycle 2 Day 7 (C2D7)) may be collected with the intention of providing further information about disease response to treatment. Depending on results of initial gene expression profiles, the timing of the biopsies may be adjusted, but without change in total number of biopsies per patient.

In a retrospective pilot study, CT scans from 20 consecutive off-study patients will be re-reviewed. Response Evaluation Criteria in Solid Tumors (RECIST) imaging measurements will be compared to volumetric density (Total Volume of Viable Tumor, TVVT) CT measurements. The objective is to establish whether volumetric density/percent necrosis algorithms such as TVVT more accurately assess extent of disease and response to therapy than standard RECIST criteria.

The total accrual ceiling is 73 participants (60 adult and 13 pediatric patients).

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have histologically confirmed alveolar soft part sarcoma. Pathology should be confirmed at the Laboratory of Pathology, National Institutes of Health.

Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 millimeters with conventional techniques or as greater than or equal to 10 millimeters with spiral computed tomography (CT) scan.

Patients must have metastatic alveolar soft part sarcoma that is not curable by surgery. Patients who have surgically resectable tumors with metastasis will be considered on a case by- case basis.

Any prior therapy must have been completed greater than or equal to 4 weeks prior to enrollment on protocol and the participant must have recovered to eligibility levels from prior toxicity. Patients should be at least 6 weeks out from nitrosoureas and mitomycin C. Prior radiation should have been completed greater than or equal to 4 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study (also referred to as an early Phase I study or pre-Phase I study where a sub-therapeutic dose of drug is administered) at the principal investigator's (PI's) discretion, and should haverecovered to eligibility levels from any toxicities.

Any degree of prior treatment is allowed, including other anti-angiogenic treatments (e.g., vascular endothelial growth factor receptor 2 (VEGFR2) inhibitors or bevacizumab). Patients with no prior therapy are eligible, provided they have metastatic disease that is not curable by surgery.

Body surface area (BSA) greater than or equal to 1.04 square meter.

Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 for adults, Karnofsky performance status greater than or equal to 50% for pediatric patients greater than 10 years of age, and Lansky performance status greater than or equal to 50 for pediatric patients less than or equal to 10 years of age.

Life expectancy of greater than 8 weeks.

Patients must have normal organ and marrow function as defined below:

* absolute neutrophil count greater than or equal to 1,500/microliter
* platelets greater than or equal to 100,000/microliter
* total bilirubin less than 1.5 times institutional upper limit of normal
* Aspartate aminotransferase (AST)(Serum glutamic Oxaloacetic transaminase (SGOT)/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase (SGPT)) less than or equal to 2.5 times institutional upper limit of normal
* creatinine within normal limits based on age as follows:

Age (Years) Maximum Serum Creatinine (milligrams per deciliter)

less than or equal to 5 0.8

5 less than age less than or equal to 10 1.0

10 less than age less than or equal to 15 1.2

greater than 15 1.5

OR

creatinine clearance greater than or equal to 60 milliliter/min for adults or greater than or equal to 60 milliliter/min/1.73m^2 for children with creatinine levels above institutional upper limit of normal.

Corrected QT interval (QTc) must be less than 500 msec.

Pediatric patients: Normal left ventricular function with ejection fraction greater than 55% or shortening fraction greater than or equal to 27%.

At present, the potential of Cediranib (AZD2171) for clinically significant drug interactions involving the cytochrome P450 (CYP) isozymes is unknown. However, studies of the agent in rats indicated possible suppression of cytochrome P450, family 1, subfamily A (CYP1A) that may be of biological significance. Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity of pharmacokinetics (PK) of AZD2171 will be determined following review of their case by the Principal Investigator. Efforts should be made to switch patients with brain metastases who are taking enzyme-inducing anticonvulsant agents to other medications one week prior to starting therapy.

AZD2171 has been shown to terminate fetal development in the rat, as expected for a process dependent on vascular endothelial growth factor (VEGF) signaling. For this reason, women of child-bearing potential must have a negative pregnancy test prior to study entry. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Ability to understand and the willingness to sign a written informed consent document.

Patients should not be receiving any other investigational agents.

Prior therapy with anti-angiogenic agents is permitted.

EXCLUSION CRITERIA:

Patients with clinically significant illnesses which would compromise participation in the study, including, but not limited to: active or uncontrolled infection, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia; or psychiatric illness/social situations that would limit compliance with study requirements.

Patients may not be receiving any medication that may markedly affect renal function (e.g., vancomycin, amphotericin, ibuprofen, pentamidine).

Patients who are unable to swallow tablets.

Mean QTc greater than 500 msec (with Bazett's correction) in screening electrocardiogram or history of familial long Q wave, T wave (QT) syndrome.

Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart.

Pregnant women are excluded from this study because AZD2171 is a VEGF inhibitor with known abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD2171, breastfeeding should be discontinued if the mother is treated with AZD2171.

Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for PK interactions with AZD2171.

Adult patients with hypertension not controlled by medical therapy (hypertension defined as systolic blood pressure greater than 150 millimeters of mercury or diastolic pressure greater than 90 millimeters of mercury despite optimal medical management). Pediatric patients must have blood pressure (BP) within normal limits (WNL) for age. NOTE: blood pressure within the upper limit of normal is defined as: blood pressure less than or equal to the 95th percentile for age, height, and gender, and measured, and not be receiving medication for treatment of hypertension.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 53 (Actual)
Dates: Start 2009-07-18 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI). Additionally, requests for all collected individual participant data (IPD) from clinical trials, conducted under a binding collaborative agreement between National Cancer Institute (NCI)/Division of Cancer Treatment and Diagnosis (DCTD) and a pharmaceutical/biotechnology company, that are not under data safety monitoring board (DSMB) monitoring must be in compliance with the terms of the binding collaborative agreement and must be approved by NCI/DCTD and the Pharmaceutical Collaborator (i.e., the NCI Experimental Therapeutics Clinical Trials Network (ETCTN) Director in conjunction with the NCI/DCTD Regulatory Affairs Branch).

REFERENCES:
- [Derived] Cohen JW, Widemann BC, Derdak J, Dombi E, Goodwin A, Dompierre J, Onukwubiri U, Steinberg SM, O'Sullivan Coyne G, Kummar S, Chen AP, Glod J. Cediranib phase-II study in children with metastatic alveolar soft-part sarcoma (ASPS). Pediatr Blood Cancer. 2019 Dec;66(12):e27987. doi: 10.1002/pbc.27987. Epub 2019 Sep 10. PMID 31502400
- [Derived] Hall PE, Shepherd STC, Brown J, Larkin J, Jones R, Ralph C, Hawkins R, Chowdhury S, Boleti E, Bahl A, Fife K, Webb A, Crabb SJ, Geldart T, Hill R, Dunlop J, McLaren D, Ackerman C, Wimalasingham A, Beltran L, Nathan P, Powles T. Radiological Response Heterogeneity Is of Prognostic Significance in Metastatic Renal Cell Carcinoma Treated with Vascular Endothelial Growth Factor-targeted Therapy. Eur Urol Focus. 2020 Sep 15;6(5):999-1005. doi: 10.1016/j.euf.2019.01.010. Epub 2019 Feb 6. PMID 30738795
- [Derived] Powles T, Brown J, Larkin J, Jones R, Ralph C, Hawkins R, Chowdhury S, Boleti E, Bhal A, Fife K, Webb A, Crabb S, Geldart T, Hill R, Dunlop J, Hall PE, McLaren D, Ackerman C, Beltran L, Nathan P. A randomized, double-blind phase II study evaluating cediranib versus cediranib and saracatinib in patients with relapsed metastatic clear-cell renal cancer (COSAK). Ann Oncol. 2016 May;27(5):880-6. doi: 10.1093/annonc/mdw014. Epub 2016 Jan 22. PMID 26802156
- [Derived] Kummar S, Allen D, Monks A, Polley EC, Hose CD, Ivy SP, Turkbey IB, Lawrence S, Kinders RJ, Choyke P, Simon R, Steinberg SM, Doroshow JH, Helman L. Cediranib for metastatic alveolar soft part sarcoma. J Clin Oncol. 2013 Jun 20;31(18):2296-302. doi: 10.1200/JCO.2012.47.4288. Epub 2013 Apr 29. PMID 23630200
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-C-0192.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult Participants w/Alveolar Soft Part Sarcoma: Adult participants will be treated with 30 mg by mouth once a day for 28 days (28-day cycles).
  AZD2171: Cediranib (AZD2171), a vascular endothelial growth factor (VEGF)/KIT tyrosine kinase inhibitor, has demonstrated antitumor activity in early phase clinical trials in adult and pediatric patients with Alveolar Soft Part Sarcoma (ASPS).
- Pediatric Participants w/Alveolar Soft Part Sarcoma: Pediatric participants (<16 years old) will be treated with 12 mg/m^2/day once a day for 28 days (28-day cycles).
  AZD2171: Cediranib (AZD2171), a vascular endothelial growth factor (VEGF)/KIT tyrosine kinase inhibitor, has demonstrated antitumor activity in early phase clinical trials in adult and pediatric patients with Alveolar Soft Part Sarcoma (ASPS).
Period: Overall Study
Arm/Group | Adult Participants w/Alveolar Soft Part Sarcoma | Pediatric Participants w/Alveolar Soft Part Sarcoma
Started | 46 | 7
Completed | 1 | 3
Not Completed | 45 | 4
Not completed — Refused further treatment | 1 | 1
Not completed — Patient was not treated | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Progressive disease | 42 | 3

BASELINE CHARACTERISTICS:
Groups:
- Pediatric Participants w/Alveolar Soft Part Sarcoma: Pediatric participants will be treated with 12 mg/m^2/day once a day for 28 days (28-day cycles).
  AZD2171: Cediranib (AZD2171), a vascular endothelial growth factor (VEGF)/KIT tyrosine kinase inhibitor, has demonstrated antitumor activity in early phase clinical trials in adult and pediatric patients with Alveolar Soft Part Sarcoma (ASPS).
- Total: Total of all reporting groups
Arm/Group | Adult Participants w/Alveolar Soft Part Sarcoma | Pediatric Participants w/Alveolar Soft Part Sarcoma | Total
Number analyzed (Participants) | 46 | 7 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 7 | 7
  Between 18 and 65 years | 46 | 0 | 46
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30 [19 to 59] | 13 [9 to 15] | 21.5 [9 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 4 | 27
  Male | 23 | 3 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 0 | 8
  Not Hispanic or Latino | 38 | 7 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 3 | 14
  White | 25 | 3 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 46 | 7 | 53
Eastern Cooperative Oncology Group (ECOG) Status [Count of Participants; unit: Participants] — ECOG status for adults indicates level of participant activity. 0 = fully active
  1. = ambulatory and can perform light work
  2. = capable of all self-care but unable to perform work activities Population: ECOG applies to the adult participants only.
  Participants
    0: number analyzed (Participants) | 46 | 0 | 46
    0 | 4 |  | 4
    1: number analyzed (Participants) | 46 | 0 | 46
    1 | 38 |  | 38
    2: number analyzed (Participants) | 46 | 0 | 46
    2 | 4 |  | 4
Lansky/Karnofsky Performance Status [Count of Participants; unit: Participants] — Lansky/Karnofsky for pediatric participants indicates level of activity. 100% = normal activity with no signs/symptoms of disease 90% = normal activity with a few signs/symptoms of disease 80% =normal activity with some difficulty Population: Lansky/Karnofsky applies to the pediatric participants only.
  Participants
    100%: number analyzed (Participants) | 0 | 7 | 7
    100% |  | 1 | 1
    90%: number analyzed (Participants) | 0 | 7 | 7
    90% |  | 4 | 4
    80%: number analyzed (Participants) | 0 | 7 | 7
    80% |  | 2 | 2
Prior Resection [Count of Participants; unit: Participants] | 35 | 3 | 38
Prior Radiation [Count of Participants; unit: Participants] | 27 | 2 | 29
Prior Systemic Therapy [Count of Participants; unit: Participants] — Population: Applies to the pediatric participants only.
  Participants
    number analyzed (Participants) | 0 | 7 | 7
    (all) |  | 4 | 4
Prior Systemic Therapies [Count of Participants; unit: Participants]
  0 | 18 | 4 | 22
  1 | 18 | 1 | 19
  2 | 5 | 0 | 5
  ≥3 | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Minimal Response Rate in Pediatric Participants With Alveolar Soft Part Sarcoma (ASPS)
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST)v1.0. A minimal response is defined as a 5% overall response rate (Partial Response (PR) + Complete Response (CR)
Time Frame: Date treatment initiated to date off study, an average of 16.9 cycles for adult patients and 34.7 cycles for pediatric patients (1 cycle = 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Participants w/Alveolar Soft Part Sarcoma
Number analyzed (Participants) | 7
Participants | 0

2. Primary Outcome: Number of Participants With a Response (Partial Response (PR) + Complete Response (CR)) of AZD2171 in Adult Participants With Alveolar Soft Part Sarcoma (ASPS)
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response is disappearance of all no-target lesions and normalization of tumor marker level. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 2 cycles (e.g., one cycle = 28 days)
Population: 45/46 participants were analyzed because one participant was not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants w/Alveolar Soft Part Sarcoma
Number analyzed (Participants) | 45
Participants
  Complete Response | 0
  Partial Response | 13

3. Primary Outcome: Number of Participants With a Best Observed Response
Description: Response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.0. Complete Response is disappearance of all target lesions and normalization of tumor marker level. Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions. Progressive disease is at least a 20% increase in the sum of the LD of target lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: Participants were followed for the duration of treatment, an average of 16.9 cycles for adult patients and 34.7 cycles for pediatric patients (1 cycle = 28 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Participants w/Alveolar Soft Part Sarcoma
Number analyzed (Participants) | 7
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 5
  Progressive Disease | 2

4. Primary Outcome: Number of Participants With a Best Response
Description: as for outcome 3
Time Frame: as for outcome 1
Population: 45/46 participants were analyzed because one participant did not receive any treatment on the trial.
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants w/Alveolar Soft Part Sarcoma
Number analyzed (Participants) | 45
Participants
  Complete Response | 0
  Partial Response | 13
  Stable Disease | 30
  Progressive Disease | 2

5. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Adult Participants w/Alveolar Soft Part Sarcoma | Pediatric Participants w/Alveolar Soft Part Sarcoma
Number analyzed (Participants) | 46 | 7
Participants | 45 | 7

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of treatment, an average of 16.9 cycles for adult patients and 34.7 cycles for pediatric patients (1 cycle = 28 days)
Arm/Group | Adult Participants w/Alveolar Soft Part Sarcoma | Pediatric Participants w/Alveolar Soft Part Sarcoma
All-Cause Mortality (participants affected / at risk) | 2/46 | 0/7
Serious Adverse Events (participants affected / at risk) | 22/46 | 6/7
Other Adverse Events (participants affected / at risk) | 45/46 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Participants w/Alveolar Soft Part Sarcoma (N=46) | Pediatric Participants w/Alveolar Soft Part Sarcoma (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CPK increased (Investigations) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Fever (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Slipped capital femoral epiphysis right side
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Death due to disease progression
Neutrophil count decreased (Investigations) | 2 (2) | 1 (2)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Papilledema (Eye disorders) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pregnancy, puerperium and perinatal conditions - Other, Pregnancy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (7) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sudden death NOS (General disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, SCFE (Surgical and medical procedures) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Testicular disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adult Participants w/Alveolar Soft Part Sarcoma (N=46) | Pediatric Participants w/Alveolar Soft Part Sarcoma (N=7)
Abdominal distension (Gastrointestinal disorders) | 3 (5) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 30 (66) | 4 (7)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 34 (130) | 3 (13)
Alkaline phosphatase increased (Investigations) | 16 (43) | 3 (15)
Allergic reaction (Immune system disorders) | 2 (2) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (9) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 18 (62) | 5 (10)
Anorexia (Metabolism and nutrition disorders) | 17 (22) | 5 (6)
Anxiety (Psychiatric disorders) | 6 (10) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 34 (126) | 3 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 14 (17) | 4 (5)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 13 (62) | 2 (35)
Blurred vision (Eye disorders) | 5 (8) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
CPK increased (Investigations) | 10 (18) | 2 (10)
Cheilitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (4)
Chills (General disorders) | 3 (7) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 13 (33) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 3 (3)
Creatinine increased (Investigations) | 7 (19) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 6 (10) | 2 (3)
Dental caries (Gastrointestinal disorders) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 5 (9) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 44 (183) | 6 (36)
Dizziness (Nervous system disorders) | 16 (26) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Ear and labyrinth disorders - Other, ear fluid collection (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema limbs (Gastrointestinal disorders) | 5 (7) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 3 (4) | 0 (0)
Endocrine disorders - Other, TSH elevated (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 (12) | 3 (10)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 1 (2) | 0 (0)
Eye disorders - Other, Retinal degeneration (Eye disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 0 (0)
Eyelid function disorder (Eye disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fatigue (General disorders) | 33 (49) | 6 (17)
Fever (General disorders) | 5 (6) | 5 (11)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (4) | 2 (2)
Flu like symptoms (General disorders) | 5 (8) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (3)
Gastrointestinal disorders - Other, Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 22 (80) | 6 (15)
Hearing impaired (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 4 (7) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 1 (2)
Hemoglobinuria (Renal and urinary disorders) | 19 (53) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hot flashes (Vascular disorders) | 3 (4) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 22 (46) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (9) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (7) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 11 (16) | 1 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 13 (15) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 35 (879) | 3 (21)
Hyperthyroidism (Endocrine disorders) | 4 (7) | 1 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 7 (23) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 27 (101) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (19) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 9 (11) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 27 (81) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 29 (71) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (28) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 33 (70) | 2 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, Total protein decreased (Immune system disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, Cold sores (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Infection in armpit (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Mouth infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other, Toe nail (Infections and infestations) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 11 (15) | 1 (1)
Investigations - Other, Bicarbonate, serum-low (Investigations) | 4 (10) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 4 (5) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 1 (4) | 0 (0)
Lung infection (Infections and infestations) | 2 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 21 (98) | 3 (20)
Malaise (General disorders) | 1 (2) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 3 (4) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 29 (51) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (3)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (18) | 1 (1)
Nausea (Gastrointestinal disorders) | 27 (56) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
Nervous system disorders - Other, Right side paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 11 (57) | 3 (54)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (8)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Otitis media (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (12) | 5 (9)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 25 (35) | 1 (3)
Palpitations (Cardiac disorders) | 4 (4) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (20) | 0 (0)
Pericardial effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 16 (71) | 4 (15)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 34 (157) | 5 (23)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 11 (19) | 2 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, Running nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis infective (Infections and infestations) | 0 (0) | 1 (1)
Scleral disorder (Eye disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Serum amylase increased (Investigations) | 1 (8) | 1 (3)
Sinus bradycardia (Cardiac disorders) | 2 (3) | 2 (2)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 5 (5) | 2 (2)
Sinusitis (Infections and infestations) | 3 (6) | 2 (3)
Skin and subcutaneous tissue disorders - Other, Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Fight laceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, Perianal irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Skin and subcut. Tissue disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6)
Stomach pain (Gastrointestinal disorders) | 2 (2) | 1 (2)
Testicular disorder (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (3) | 2 (2)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (22) | 2 (5)
Upper respiratory infection (Infections and infestations) | 10 (10) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 11 (13) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (2) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 3 (3) | 0 (0)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Vascular disorders - Other, Hemoptysis (Vascular disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 1 (1)
Vomiting (Gastrointestinal disorders) | 23 (67) | 4 (5)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Weight gain (Investigations) | 2 (3) | 0 (0)
Weight loss (Investigations) | 25 (78) | 3 (9)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 22 (79) | 3 (40)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Lymphocyte count increased (Investigations) | 3 (4) | 0 (0)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thyroid stimulating hormone increased (Investigations) | 0 (0) | 2 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Immune system disorders - Other, Left inguinal adenopathy (Immune system disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, callouses on both feet (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/77/NCT00942877/Prot_SAP_002.pdf
  • Informed Consent Form (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT00942877/ICF_003.pdf